CLINICAL TRIAL: NCT00476905
Title: Spectral Diagnosis of Cutaneous Malignancy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0856
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Skin Cancer
Keywords: Basal Cell Carcinoma; Squamous Cell Carcinoma; Pre-Cancer Lesions; Pigmented Lesions; Benign Lesions; Skin Cancer; Spectral Diagnosis; Optical Spectroscopy
MeSH Terms: conditions — Skin Neoplasms; Carcinoma, Basal Cell; Carcinoma, Squamous Cell | interventions — Spectrum Analysis, Raman

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spectral-Diagnosis: Method for noninvasive detection of cutaneous malignancies
  Interventions: Device: Spectral Diagnosis Probe

INTERVENTIONS:
Device: Spectral Diagnosis Probe — The device collects two types of tissue spectra: i) laser-induced fluorescence spectra and ii) white light reflectance spectra. This portable reflectance spectrofluorimeter collects spectra in a fraction of a second. Light collection and delivery are achieved via an optical fiber probe. The optical fiber probe is approximately 1 mm in diameter and 3 m long. The same probe collects light emitted from the tissue and delivers it back to the instrument for spectral analysis.
  Other Names: Optical Spectroscopy

SUMMARY:
The goal of this clinical research study is to evaluate the use of an imaging technology called spectral diagnosis. Researchers want to find out if a special spectral-diagnosis probe can be used to detect skin cancers.

DETAILED DESCRIPTION:
The spectral-diagnosis probe being used in this study uses dim pulses of light to identify features of tissue that may be related to the status of skin cancer. The probe is shaped like a catheter, and it has a camera on the end, which takes pictures of the skin.

If you agree to take part in this study, you will be asked questions about your age, race, smoking status, and the status of any diseases you may have (such as diabetes, connective tissue disease, and infectious disease). It should take about 5 minutes to answer these questions.

The study doctor will then decide which of your lesions are suitable for imaging by the probe. If necessary, any hair on or around the lesion(s) will be shaved or trimmed. The area(s) of skin being imaged will be cleaned with rubbing alcohol.

As part of your exam, the study doctor will use the probe to measure the selected areas of tissue. To perform the spectral-diagnosis measurement, the probe will be gently placed on the surface of your skin. Each selected area of your skin will take about a few seconds to image. The probe will shine different types of light onto the skin, and it will collect the light that reflects from the skin surface. The light signals will be stored so that researchers can look at them. Preparing the lesion, imaging it, and collecting the light signals should take about 10-15 minutes per lesion.

After all of the imaging is over, you will have biopsies performed on the lesions that your study doctor has decided are in need of such treatment as part of your standard care.

After this clinic visit, your participation in the study will be over.

This is an investigational study. The imaging probe is not commercially available or FDA approved. At this time, it is being used in research only. Up to 150 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female and over 18 years of age.
2. Patients undergoing an examination of their skin
3. Patients with a lesion(s) in one of the five categories: basal cell carcinoma, squamous cell carcinoma, pre-cancer lesions, pigmented lesions, and benign lesions
4. Patients whose lesion also warrants a biopsy.
5. Signed informed consent document.

Exclusion Criteria:

1. Patients with absence of skin lesion(s) in one of the five categories.
2. Patients whose identified lesion did not need a biopsy.
3. Patients who did not sign the informed consent and agree to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, at routine skin examination, found to have a lesion(s) in one of the five categories: basal cell carcinoma, squamous cell carcinoma, pre-cancer lesions, pigmented lesions, and benign lesions, which may also warrant biopsy.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2007-04 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Spectroscopic features of skin lesions in vivo | Preparing lesion, imaging it, and collecting the light signals should take about 10-15 minutes per lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Migden, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org